CLINICAL TRIAL: NCT00973076
Title: A Phase I, Open Label, Single-centre Study to Assess the Safety and Tolerability of the Tor Kinase Inhibitor AZD8055 Administered Orally to Japanese Patients With Advanced Solid Tumours
Brief Title: Study to Assess the Safety and Tolerability of the Tor Kinase Inhibitor AZD8055
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1600C00003
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Cancer; Solid Tumors; Advanced Solid Malignancies
Keywords: Phase I, cancer; solid tumors; advanced solid malignancies; dose escalation; mTOR Kinase Inhibitor; Japanese
MeSH Terms: conditions — Neoplasms | interventions — (5-(2,4-bis((3S)-3-methylmorpholin-4-yl)pyrido(2,3-d)pyrimidin-7-yl)-2-methoxyphenyl)methanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD8055 (Experimental): AZD8055 will be administered orally
  Interventions: Drug: AZD8055

INTERVENTIONS:
Drug: AZD8055 — Tablets, orally administered, twice daily

SUMMARY:
The primary objective is to assess the safety and tolerability of AZD8055 in Japanese patients with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with advanced solid tumors for which suitable effective standard treatment does not exist or is no longer effective
* Relatively good overall health other than cancer

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells)
* Poor liver or kidney function
* Serious concomitant illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events, clinical laboratory tests (clinical chemistry, haematology, coagulation, urinalysis), glucose management (s-glucose, s-insulin, haemoglobin A1c [HbA1c]), vital signs (pulse rate, blood pressure, weight and body temperature) | Laboratory values, vital sign, physical examination every week during Cycle 1 and 2.

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of AZD8055 following both single and multiple oral dosing in patients with advanced solid tumours | According to protocol specified schedule, the number of PK samples collected during Cycle 1
To seek preliminary evidence of the anti-tumour activity of AZD8055 in patients with advanced solid malignancies as measured by objective tumour response (according to RECIST criteria) | Every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, Study Director — AstraZeneca; Tomohide Tamura, Principal Investigator — National Cancer Center Hospital
Locations (1):
- Research Site, Tokyo, Japan

REFERENCES:
- [Derived] Asahina H, Nokihara H, Yamamoto N, Yamada Y, Tamura Y, Honda K, Seki Y, Tanabe Y, Shimada H, Shi X, Tamura T. Safety and tolerability of AZD8055 in Japanese patients with advanced solid tumors; a dose-finding phase I study. Invest New Drugs. 2013 Jun;31(3):677-84. doi: 10.1007/s10637-012-9860-4. Epub 2012 Jul 28. PMID 22843211